CLINICAL TRIAL: NCT00963651
Title: GE Healthcare VolumeRAD Lung Nodule Detection Study
Status: Completed | Type: Observational
Sponsor: American College of Radiology - Image Metrix (Industry)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: GE-VORTEX; GE 2901
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Pulmonary Nodule, Solitary; Multiple Pulmonary Nodules
Keywords: Pulmonary nodule, solitary; Multiple pulmonary nodules
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspicion of pulmonary nodules: Eligible participants will include those referred for x-ray computed tomography (CT) of the chest for suspicion of a pulmonary nodule or other unrelated reasons.
  Interventions: Device: Chest tomosynthesis and X-ray

INTERVENTIONS:
Device: Chest tomosynthesis and X-ray — VolumeRAD tomosynthesis; Conventional Chest X-ray; Dual energy (bone and soft tissue PA chest images)

SUMMARY:
To perform a multiple reader, multiple case (MRMC) observer study assessing the detection performance of VolumeRAD tomosynthesis of the chest in detecting lung nodules.

DETAILED DESCRIPTION:
Digital tomosynthesis is a form of limited angle tomography that creates a series of section images using a conventional x-ray tube and generator, a digital detector, and appropriate reconstruction software. It creates section images from a series of projection images acquired as the x-ray tube moves along a prescribed path. Because tomosynthesis can minimize the visual presence of overlying anatomy - the ribs, for example - it has the potential to improve the detection of lesions such as pulmonary nodules when compared with conventional chest radiography.

The primary aim of this study is to determine whether the use of VolumeRAD tomosynthesis, in addition to CxR, increases physician accuracy in the detection of lung nodules between 3mm and 20mm in diameter when compared to conventional posterior-anterior (PA) and lateral (LAT) chest radiography (CxR). This aim will be addressed by measuring free-response performance of experienced (with VolumeRAD), blinded expert readers' detection performance. Specifically, we will compare detection performance, as measured by the area under the alternative free response receiver operating characteristic (AFROC) curve, among readers viewing PA and LAT chest X-rays versus VolumeRAD tomosynthesis. The nodule will be the unit of analysis.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for chest CT as part of their needed medical care;
* If available, individuals who have had previous imaging to suggest they fulfill the needs of the study;
* 18 years of age, or older;
* In good enough physical condition to stand motionless and hold their breath during the image acquisition procedures.

Exclusion Criteria:

* Children under 18 years of age;
* Women who are pregnant or who suspect they may be pregnant;
* Individuals who on previous imaging are shown to have objects in or around the lungs that might produce substantial artifacts that would obscure pulmonary nodules;
* Individuals who on recent imaging had active lung or pleural disease that would obscure pulmonary nodules;
* Individuals with more than 5 pulmonary nodules between 5mm and 20mm in diameter in either right or left lung.
* Individuals suspected to have more than 15 total nodules between 3mm and 20mm. NOTE that up to 20 nodules between 3mm and 20mm will be allowed in the final study sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include those referred for x-ray computed tomography (CT) of the chest for suspicion of a pulmonary nodule or other unrelated reasons.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2009-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Multi-reader, multi-case Receiver Operating Characteristics (ROC) methodology. | Post accrual of 210 participants
  The primary objective of this study is to determine if the use of VolumeRAD tomosynthesis increases the accuracy of the detection of lung nodules between 3mm and 20mm in diameter when compared to conventional PA and lateral chest radiography alone.

SECONDARY OUTCOMES:
Actionability classification accuracy of all modalities | Multipe reader, multiple case reader study

CONTACTS AND LOCATIONS:
Overall Officials: James Dobbins, MD, Principal Investigator — Duke University
Locations (4):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - University of Washington Medical Center, Seattle, Washington
- Sahlgrenska University Hospital, Gothenburg, Sweden